CLINICAL TRIAL: NCT01057693
Title: A PHASE 3B MULTICENTER, DOUBLE-BLIND, RANDOMIZED WITHDRAWAL EFFICACY AND SAFETY STUDY OF PREGABALIN IN THE TREATMENT OF PATIENTS WITH INADEQUATELY TREATED PAINFUL DIABETIC PERIPHERAL NEUROPATHY
Brief Title: Study Of Pregabalin (Lyrica) In Patients With Painful Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A0081242; 2009-017389-21 (EudraCT Number)
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Results first posted 2013-02-22 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2019-02

CONDITIONS: Diabetic Neuropathy, Painful
Keywords: Diabetic peripheral neuropathy; Lyrica; pregabalin; pain
MeSH Terms: conditions — Diabetic Neuropathies; Pain | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- pregabalin (Lyrica) (Experimental)
  Interventions: Drug: pregabalin (Lyrica)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: pregabalin (Lyrica) — Lyrica 150-300 mg/day. Medication is supplied as capsules and given 3 times daily.
  Arms: pregabalin (Lyrica)
Drug: Placebo — Placebo is supplied as capsules and given 3 times daily.
  Arms: Placebo

SUMMARY:
Patients will be switched from their current medication for painful diabetic peripheral neuropathy to evaluate the safety and efficacy of pregabalin as compared to placebo. All patients will receive pregabalin, and half of patients will receive placebo at some point during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have painful diabetic peripheral neuropathy and be receiving treatment for this condition.

Exclusion Criteria:

* Patients with other pain conditions cannot participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 633 (Actual)
Dates: Start 2010-03-31 (Actual); Primary Completion 2012-01-30 (Actual); Study Completion 2012-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (171):
- United States (150):
  - Greystone Medical Research, LLC, Birmingham, Alabama
  - Neurology Clinic, PC, Northport, Alabama
  - Horizon Clinical Research Associates, PLLC, Gilbert, Arizona
  - Dedicated Clinical Research, Inc., Goodyear, Arizona
  - Dedicated Clinical Research, Goodyear, Arizona
  - Novara Clinical Research, Mesa, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Radiant Research, Inc., Scottsdale, Arizona
  - Genova Clinical Research, Inc., Tucson, Arizona
  - Central Arkansas Research, Hot Springs, Arkansas
  - Little Rock Diagnostic Clinic, Little Rock, Arkansas
  - Convergys Clinical Research, Inc., Anaheim, California
  - Providence Clinical Research, Burbank, California
  - Valley Research, Fresno, California
  - Center for United Research, Inc., Lakewood, California
  - Healthcare Partners Medical Group, Los Angeles, California
  - University of Southern California, Keck School of Medicine, Department of Neurology, Los Angeles, California
  - Richard S. Cherlin, MD, Los Gatos, California
  - Northridge Neurological Research, Northridge, California
  - Remek Research, Pomona, California
  - Sierra Clinical Research, Roseville, California
  - CNRI-San Diego, LLC, San Diego, California
  - San Diego Clinical Trials, San Diego, California
  - Center for Clinical Research, Inc., San Francisco, California
  - Apex Research Institute, Santa Ana, California
  - Neurological Research Institute, Santa Monica, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Foothills Pain Management, West Covina, California
  - Aurora Family Medicine Center, PC, Aurora, Colorado
  - Alpine Clinical Research Center, Inc., Boulder, Colorado
  - Mountain View Clinical Research, Denver, Colorado
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Metabolic Research Institute, Inc., Boynton Beach, Florida
  - Bradenton Research Center, Bradenton, Florida
  - Meridien Research, Bradenton, Florida
  - Meridien Research, Brooksville, Florida
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Deerfield Beach Cardiology Research, Deerfield Beach, Florida
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - MD Clinical, Hallandale, Florida
  - Elite Research Institute, Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Laszlo J. Mate, MD, North Palm Beach, Florida
  - Family Care Specialists, Inc., Ocala, Florida
  - Renstar Medical Research, Ocala, Florida
  - Compass Research, LLC, Orlando, Florida
  - Palm Beach Neurological Center, Advanced Research Consultants, Inc., Palm Beach Gardens, Florida
  - Suncoast Clinical Research, Palm Harbor, Florida
  - Meridien Research, St. Petersburg, Florida
  - Neurology Clinical Research, Inc., Sunrise, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Meridien Research, Tampa, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - NeuroTrials Research, Incorporated, Atlanta, Georgia
  - CPM Research Institute, Austell, Georgia
  - Columbus Research Foundation, Columbus, Georgia
  - Rockdale Medical Research Associates, Conyers, Georgia
  - Prism Research Group, Rome, Georgia
  - Valley Health Care, Rome, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Advanced Clinical Research, Meridian, Idaho
  - AMR Sakeena Research, Aurora, Illinois
  - Chicago Research Center, Inc., Chicago, Illinois
  - American Medical Research, Inc., Oak Brook, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - American Health Network, Greenfield, Indiana
  - Rehabilitation Associates of Indiana, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Kentucky Medical Research Center, Lexington, Kentucky
  - Endocrinology Center of Southwest Louisiana, Lake Charles, Louisiana
  - Heartland Research, LLC, Lake Charles, Louisiana
  - Primary Physician Care, LLC, Lake Charles, Louisiana
  - Arthritis and Diabetes Clinic, Inc, Monroe, Louisiana
  - Miray Medical Center, Brockton, Massachusetts
  - Clinical Research Center of Cape Cod, Inc., Hyannis, Massachusetts
  - MedVadis Research Corporation, Watertown, Massachusetts
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - Harris and Associates MD, PC, Detroit, Michigan
  - Borgess Diabetes Center, Kalamazoo, Michigan
  - Borgess Research Institute, Kalamazoo, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - KMED Research, Saint Clair Shores, Michigan
  - William Beaumont Hospital, Troy, Michigan
  - Troy Internal Medicine, PC, Troy, Michigan
  - MAPS Applied Research Center, Inc., Edina, Minnesota
  - Medical Advanced Pain Specialists (MAPS), Edina, Minnesota
  - Medical Advanced Pain Specialists, Maple Grove, Minnesota
  - Medical Advanced Pain Specialists, Shakopee, Minnesota
  - CRC of Jackson, Jackson, Mississippi
  - Physician's Surgery Center, Jackson, Mississippi
  - Randall T. Huling, Jr., MD, CPI, Olive Branch, Mississippi
  - University of Missouri Healthcare/Cosmopolitan Diabetes and Endocrinology Center, Columbia, Missouri
  - Melinda A. Crockett-Maples, Marionville, Missouri
  - Clinvest, Springfield, Missouri
  - A & A Pain Institute of Saint Louis, St Louis, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Lincoln Internal Medicine Associates, Lincoln, Nebraska
  - Desert Endocrinology Clinical Research Center, Henderson, Nevada
  - Desert Endocrinology, Las Vegas, Nevada
  - Office of Dr. Danka Michaels, MD, Las Vegas, Nevada
  - Office of Stephen Miller, M.D., Las Vegas, Nevada
  - Raleigh Neurology Associates, P.A., Raleigh, North Carolina
  - Carolina Pharmaceutical Research, Statesville, North Carolina
  - Radiant Research, Inc., Akron, Ohio
  - Community Research, Cincinnati, Ohio
  - Radiant Research, Cincinnati, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - Providence Health Partners - Center for Clinical Research, Dayton, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Veronique Sebastian, MD, Oklahoma City, Oklahoma
  - Angelique Barreto, MD, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Blair Orthopedic Associates, Inc., Altoona, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Research Protocol Management Specialists, Pittsburgh, Pennsylvania
  - Coastal Medical, East Greenwich, Rhode Island
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Omega Medical Research, Warwick, Rhode Island
  - Aiken Center for Clinical Research, Aiken, South Carolina
  - TLM Medical Services, LLC, Columbia, South Carolina
  - Radiant Research Inc., Greer, South Carolina
  - Neurology and Pain Clinic, LLC, Orangeburg, South Carolina
  - University Diabetes & Endocrine Consultants, Chattanooga, Tennessee
  - SCRI Research Center, Germantown, Tennessee
  - Sarah Cannon Research Institute, Jackson, Tennessee
  - AM Diabetes & Endocrinology Center, Memphis, Tennessee
  - Memphis Internal Medicine, Memphis, Tennessee
  - ClinRx Research LLC, Carrollton, Texas
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Medical Group of Texas, Fort Worth, Texas
  - The Nerve and Muscle Center of Texas, Houston, Texas
  - ClinRx Research, LLC, Richardson, Texas
  - Paragon Research Center, LLC, San Antonio, Texas
  - Alamo Clinical Research, San Antonio, Texas
  - Cetero Research - San Antonio, San Antonio, Texas
  - Pioneer Research Solutions, Inc, Sugar Land, Texas
  - L. Craig Larsen and Clark C. Larsen, Murray, Utah
  - Aspen Clinical Research, Orem, Utah
  - Daniel B. Vine, MD, Salt Lake City, Utah
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Jean Brown Research, Salt Lake City, Utah
  - Foot and Ankle Clinic, West Jordan, Utah
  - Neurological Associates, Incorporated, Henrico, Virginia
  - National Clinical Research - Norfolk, Inc., Norfolk, Virginia
  - Spokane Internal Medicine, Spokane, Washington
  - Aurora Advanced Healthcare, Inc., Milwaukee, Wisconsin
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - Winnipeg Health Sciences Centre, Winnipeg, Manitoba
  - Winnipeg Regional Health Authority Sciences Centre Winnipeg, Winnipeg, Manitoba
  - Capital District Health Authority, QEII Health Sciences Centre, Halifax, Nova Scotia
  - The Ottawa Hospital, Riverside Campus - Riverside Professional Building, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
- Puerto Rico (2):
  - Ponce School of Medicine & Health Sciences, Ponce
  - Instituto de Endocrinologia Diabetes y Metabolismo, Toa Baja
- South Africa (13):
  - Bloemfontein Medi-Clinic, Bloemfontein, Free State
  - Dr Makan's Rooms, Johannesburg, Gauteng
  - Chris Hani Baragwanath Hospital, Soweto, Gauteng
  - Randles Road Medical Centre, Durban, KwaZulu-Natal
  - Chelmsford Medical Centre, Durban, KwaZulu-Natal
  - Centre for Diabetes and Endocrinology, Durban, KwaZulu-Natal
  - Dr Jeevren Reddy's Surgery, KwaDukuza, KwaZulu-Natal
  - Parklands Medical Centre, Overport, KwaZulu-Natal
  - Dot Shuttleworth Centre for Diabetes, Durban, Overport
  - Centre for Diabetes and Endocrinology, Houghton, Johannesburg
  - 102 Parklands Medical Centre, Overport, Durban
  - Dr's Sauermann and Meyer, Polokwane
  - Diabetes Care Centre, Pretoria

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Raskin P, Huffman C, Toth C, Asmus MJ, Messig M, Sanchez RJ, Pauer L. Pregabalin in patients with inadequately treated painful diabetic peripheral neuropathy: a randomized withdrawal trial. Clin J Pain. 2014 May;30(5):379-90. doi: 10.1097/AJP.0b013e31829ea1a1. PMID 23887339
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081242&StudyName=Study%20Of%20Pregabalin%20%28Lyrica%29%20In%20Patients%20With%20Painful%20Diabetic%20Peripheral%20Neuropathy

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregabalin SB: Participants who were inadequately controlled on their current diabetic peripheral neuropathy (DPN) treatment were switched to single-blind (SB) pregabalin capsules at a starting dose of 150 milligram per day (mg/day) and increased to 300 mg/day, administered three times daily up to Week 6. Participants who experienced greater than or equal to (>=) 30 percent (%) pain reduction from baseline to Week 6 were eligible for double-blind (DB) treatment phase.
- Pregabalin DB: Participants who experienced >=30% pain reduction in SB treatment phase, after Week 6 received pregabalin capsules 150 mg/day or 300 mg/day, administered three times daily up to Week 19 during DB treatment phase.
- Placebo: Participants who experienced >=30% pain reduction in SB treatment phase, after Week 6 received matching placebo capsules, administered three times daily up to Week 19 during DB treatment phase.
Period: Single-Blind Phase (Up to Week 6)
Arm/Group | Pregabalin SB | Pregabalin DB | Placebo
Started | 665 | 0 | 0
Completed | 566 | 0 | 0
Not Completed | 99 | 0 | 0
Not completed — Adverse Event | 45 | 0 | 0
Not completed — Lack of Efficacy | 7 | 0 | 0
Not completed — Lost to Follow-up | 14 | 0 | 0
Not completed — Protocol Violation | 9 | 0 | 0
Not completed — Withdrawal by Subject | 22 | 0 | 0
Not completed — Other | 2 | 0 | 0
Period: Between Single-Blind and Double-Blind
Arm/Group | Pregabalin SB | Pregabalin DB | Placebo
Started | 566 | 0 | 0
Completed | 296 | 0 | 0
Not Completed | 270 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0
Not completed — Lack of Efficacy | 247 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Protocol Violation | 7 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0
Not completed — Other | 6 | 0 | 0
Period: Double-Blind Phase (Week 7 to Week 19)
Arm/Group | Pregabalin SB | Pregabalin DB | Placebo
Started | 0 | 147 | 149
Treated | 0 | 147 | 147
Completed | 0 | 125 | 113
Not Completed | 0 | 22 | 36
Not completed — Adverse Event | 0 | 8 | 11
Not completed — Lack of Efficacy | 0 | 3 | 8
Not completed — Lost to Follow-up | 0 | 2 | 5
Not completed — Protocol Violation | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 8 | 6
Not completed — Other | 0 | 1 | 0
Not completed — Randomized, Not Treated | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Pregabalin SB: Participants who were inadequately controlled on their current DPN treatment were switched to SB pregabalin capsules at a starting dose of 150 mg/day and increased to 300 mg/day, administered three times daily up to Week 6. Participants who experienced >=30% pain reduction from baseline to Week 6 were eligible for DB treatment phase.
Arm/Group | Pregabalin SB
Number analyzed (Participants) | 665
Age, Customized [Number; unit: participants]
  18 to 44 Years | 58
  45 to 64 Years | 417
  >=65 Years | 190
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 302
  Male | 363

OUTCOME MEASURES:

1. Primary Outcome: Change From Single-Blind Baseline in Mean Pain Score at Week 19 During Double-Blind Phase
Description: Mean pain score was defined as the mean of the last 7 daily diary pain ratings. Participants rated their DPN pain over the past 24 hours on an 11-point numeric rating scale ranging from 0 = no pain to 10 = worst possible pain. A rating of 1-3 was considered as mild pain; 4-6 = moderate pain; and 7-10 = severe pain. SB baseline refers to the last 7 pain diary entries up to and including Day 1.
Time Frame: SB Baseline, Week 19 (DB Phase)
Population: Full analysis set (FAS) included all participants randomized to double-blind treatment who received at least 1 dose of double-blind study treatment. Missing data were imputed using Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin DB | Placebo
Number analyzed (Participants) | 147 | 147
units on a scale
  Single-Blind Baseline | 6.8 (1.24) | 6.7 (1.32)
  Change at Week 19 (DB Phase) | -3.9 (1.92) | -3.5 (2.10)
Statistical Analysis 1: Comparison: Pregabalin DB vs Placebo; P-value was calculated using analysis of covariance (ANCOVA), with terms for baseline mean pain score, center and treatment in the model; Test type: Superiority or Other; p = 0.1221, ANCOVA; Least Squares Mean Difference = -0.32, 95% CI 2-sided [-0.74 to 0.09]

2. Secondary Outcome: Time to Loss of Pain Response (Double-Blind Phase)
Description: Time to loss of pain response (based on the daily pain diary data) during the DB treatment phase was analyzed using survival analysis technique. Loss of pain response was defined as less than (<) 15% pain response relative to the SB baseline. SB baseline refers to the last 7 pain diary entries up to and including Day 1.
Time Frame: SB Baseline up to Week 19
Population: FAS included all participants randomized to double-blind treatment who received at least 1 dose of double-blind study treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pregabalin DB | Placebo
Number analyzed (Participants) | 147 | 147
days | NA [NA to NA] — Median and 95% confidence interval (CI) were not estimable because less than 50% participants experienced loss of pain response. | NA [NA to NA] — Median and 95% confidence interval (CI) were not estimable because less than 50% participants experienced loss of pain response.

3. Secondary Outcome: Change From Single-Blind Baseline in Mean Pain Score at Week 6 During Single-Blind Phase
Description: as for outcome 1
Time Frame: SB Baseline, Week 6 (SB Phase)
Population: Single-Blind Analysis Set (SBAS) included all participants who were enrolled in single-blind treatment phase and received at least 1 dose of study treatment. "N" (number of participants analyzed): participants who were evaluable for this measure and "n": participants who were evaluable for specified time-point. Missing data were imputed using LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin SB
Number analyzed (Participants) | 663
units on a scale
  SB Baseline (n= 663) | 6.7 (1.27)
  Change at Week 6 (SB Phase) (n= 658) | -2.2 (2.03)

4. Secondary Outcome: Weekly Mean Pain Scores (Single-Blind Phase)
Description: Weekly mean pain score was defined as the mean of the daily diary pain ratings split into 7 day intervals. Participants rated their DPN pain over the past 24 hours on an 11-point numeric rating scale ranging from 0 = no pain to 10 = worst possible pain. A rating of 1-3 was considered as mild pain; 4-6 = moderate pain; and 7-10 = severe pain.
Time Frame: Week 1, 2, 3, 4, 5, 6
Population: SBAS included all participants who were enrolled in single-blind treatment phase and received at least one dose of study treatment. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure and "n" signifies participants who were evaluable for specified time-point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin SB
Number analyzed (Participants) | 657
units on a scale
  Week 1 (n= 657) | 6.0 (1.62)
  Week 2 (n= 636) | 5.4 (1.82)
  Week 3 (n= 613) | 4.9 (1.93)
  Week 4 (n= 585) | 4.6 (1.93)
  Week 5 (n= 565) | 4.5 (1.92)
  Week 6 (n= 548) | 4.3 (2.02)

5. Secondary Outcome: Weekly Mean Pain Scores (Double-Blind Phase)
Description: Weekly mean pain score was defined as the mean of the daily diary pain ratings split into 7 day intervals. Participants rated their DPN pain over the past 24 hours on an 11-point numeric rating scale ranging from 0 = no pain to 10 = worst possible pain. A rating of 1-3 was considered as mild pain; 4-6 = moderate pain; and 7-10 = severe pain. SB baseline refers to the last 7 pain diary entries up to and including Day 1. DB baseline refers to the last 7 pain diary entries up to and including DB Day 1.
Time Frame: DB Baseline, Week 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19
Population: FAS included all participants randomized to double-blind treatment who received at least 1 dose of double-blind study treatment. Here "n" signifies participants who were evaluable for specified time-point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin DB | Placebo
Number analyzed (Participants) | 147 | 147
units on a scale
  DB Baseline (n= 147, 147) | 3.1 (1.42) | 3.0 (1.40)
  Week 7 (n= 144, 145) | 3.2 (1.60) | 3.3 (1.80)
  Week 8 (n= 143, 142) | 3.2 (1.72) | 3.6 (1.79)
  Week 9 (n= 140, 133) | 3.0 (1.65) | 3.4 (1.76)
  Week 10 (n= 138, 133) | 3.0 (1.70) | 3.4 (1.77)
  Week 11 (n= 138, 128) | 2.9 (1.64) | 3.3 (1.63)
  Week 12 (n= 135, 123) | 2.9 (1.68) | 3.2 (1.70)
  Week 13 (n= 134, 122) | 2.9 (1.68) | 3.1 (1.69)
  Week 14 (n= 133, 122) | 2.9 (1.64) | 3.1 (1.70)
  Week 15 (n= 131, 118) | 2.9 (1.63) | 3.0 (1.64)
  Week 16 (n= 132, 118) | 2.8 (1.65) | 3.0 (1.58)
  Week 17 (n= 128, 115) | 2.7 (1.61) | 2.9 (1.70)
  Week 18 (n= 128, 115) | 2.8 (1.66) | 2.9 (1.73)
  Week 19 (n= 115, 104) | 2.7 (1.57) | 2.8 (1.71)

6. Secondary Outcome: Percentage of Participants With At Least 30 Percent and 50 Percent Reduction in Mean Pain Score (Single-Blind Phase)
Description: Mean pain score was defined as the mean of the last 7 daily diary pain ratings. Participants rated their DPN pain over the past 24 hours on an 11-point numeric rating scale ranging from 0 = no pain to 10 = worst possible pain. A rating of 1-3 was considered as mild pain; 4-6 = moderate pain; and 7-10 = severe pain. Percentage of participants who had at least 30% and 50% pain reduction from SB baseline to Week 6 is reported. SB baseline refers to the last 7 pain diary entries up to and including Day 1.
Time Frame: Week 6
Population: SBAS included all participants who were enrolled into the single-blind treatment phase and received at least 1 dose of study treatment. Missing data were imputed using LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin SB
Number analyzed (Participants) | 665
percentage of participants
  >=30 % Reduction | 49.92
  >=50 % Reduction | 27.22

7. Secondary Outcome: Percentage of Participants With At Least 30 Percent and 50 Percent Reduction in Mean Pain Score (Double-Blind Phase)
Description: Mean pain score was defined as the mean of the last 7 daily diary pain ratings. Participants rated their DPN pain over the past 24 hours on an 11-point numeric rating scale ranging from 0 = no pain to 10 = worst possible pain. A rating of 1-3 was considered as mild pain; 4-6 = moderate pain; and 7-10 = severe pain. Percentage of participants who had at least 30% and 50% pain reduction from SB baseline to Week 19 is reported.
Time Frame: Week 19
Population: FAS included all participants randomized to double-blind treatment who received at least 1 dose of double-blind study treatment. Missing data were imputed using LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin DB | Placebo
Number analyzed (Participants) | 147 | 147
percentage of participants
  >=30% Reduction | 82.99 | 79.19
  >=50% Reduction | 62.59 | 55.03

8. Secondary Outcome: Patient Global Impression of Change (PGIC) (Single-Blind Phase)
Description: PGIC: participant rated instrument to measure participant's change in overall status on a 7-point scale; range from 1 (very much improved) to 7 (very much worse). Number of participants in each category are reported.
Time Frame: Week 6
Population: SBAS included all participants who were enrolled into the single-blind treatment phase and received at least one dose of study treatment. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Pregabalin SB
Number analyzed (Participants) | 620
participants
  Very Much Improved | 93
  Much Improved | 221
  Minimally Improved | 194
  No Change | 65
  Minimally Worse | 29
  Much Worse | 15
  Very Much Worse | 3

9. Secondary Outcome: Patient Global Impression of Change (PGIC) (Double-Blind Phase)
Description: as for outcome 8
Time Frame: Week 19
Population: FAS included all participants randomized to double-blind treatment who received at least 1 dose of double-blind study treatment. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Pregabalin DB | Placebo
Number analyzed (Participants) | 138 | 134
participants
  Very Much Improved | 23 | 23
  Much Improved | 50 | 46
  Minimally Improved | 27 | 28
  No Change | 28 | 20
  Minimally Worse | 9 | 6
  Much Worse | 1 | 8
  Very Much Worse | 0 | 3

10. Secondary Outcome: Medical Outcomes Study -Sleep Scale (MOS-SS) (Single-Blind Phase)
Description: Participant-rated 12-item questionnaire to assess constructs of sleep over past week; 7 subscales: sleep disturbance (range 0-100), snoring (range 0-100), awaken short of breath (SOB) or with headache (range 0-100), sleep adequacy (range 0-100), somnolence (range: 0-100); sleep quantity (range: 0-24), optimal sleep (yes/no), and 9 item index measures of sleep disturbance provide composite scores: sleep problems index (range 0-100). Except adequacy, optimal sleep and quantity, higher scores=more impairment.
Time Frame: SB Baseline, Week 6
Population: SBAS included all participants who were enrolled into the single-blind treatment phase and received at least one dose of study medication. Here "n" signifies participants who were evaluable for specified time-point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin SB
Number analyzed (Participants) | 665
units on a scale
  SB Baseline: Sleep disturbance (n= 665) | 53.6 (24.00)
  SB Baseline: Snoring (n= 664) | 44.7 (34.73)
  SB Baseline: Awaken SOB or With Headache (n=665) | 18.9 (24.18)
  SB Baseline: Quantity of sleep (n=663) | 5.9 (1.40)
  SB Baseline: Sleep Adequacy (n=665) | 39.2 (23.22)
  SB Baseline: Somnolence (n=665) | 42.6 (23.49)
  SB Baseline: Sleep Problems Index (n=665) | 49.2 (18.17)
  Week 6: Sleep disturbance (n= 621) | 33.6 (24.31)
  Week 6: Snoring (n= 621) | 39.9 (34.83)
  Week 6: Awaken SOB or With Headache (n= 621) | 12.6 (22.64)
  Week 6: Quantity of sleep (n= 615) | 6.6 (1.64)
  Week 6: Sleep Adequacy (n= 621) | 52.6 (25.55)
  Week 6: Somnolence (n= 621) | 34.2 (24.11)
  Week 6: Sleep Problems Index (n= 621) | 34.4 (18.82)

11. Secondary Outcome: Medical Outcomes Study -Sleep Scale (MOS-SS) (Double-Blind Phase)
Description: as for outcome 10
Time Frame: Week 19
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin DB | Placebo
Number analyzed (Participants) | 138 | 134
units on a scale
  Sleep disturbance | 26.6 (21.69) | 30.9 (23.05)
  Snoring | 41.9 (36.24) | 35.4 (35.95)
  Awaken SOB or With Headache | 12.3 (23.72) | 12.2 (23.89)
  Quantity of sleep | 6.7 (1.34) | 6.5 (1.47)
  Sleep Adequacy | 59.2 (28.67) | 59.0 (27.67)
  Somnolence | 29.7 (24.39) | 30.6 (22.98)
  Sleep Problems Index | 28.5 (17.86) | 30.9 (18.59)

12. Secondary Outcome: Number of Participants With Optimal Sleep Assessed Using Medical Outcomes Study-Sleep Scale (MOS-SS) (Single-Blind Phase)
Description: MOS-SS: participant-rated 12 item questionnaire to assess constructs of sleep over past week. It included 7 subscales: sleep disturbance, snoring, awaken short of breath or with headache, sleep adequacy, somnolence, sleep quantity, optimal sleep, and 9 item index measures of sleep disturbance provide composite scores: sleep problems index. Participants responded whether their sleep was optimal or not optimal by choosing yes or no.
Time Frame: SB Baseline, Week 6
Population: SBAS included all participants who were enrolled into the single-blind treatment phase and received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Pregabalin SB
Number analyzed (Participants) | 665
participants
  SB Baseline | 180
  Week 6 | 266

13. Secondary Outcome: Number of Participants With Optimal Sleep Assessed Using Medical Outcomes Study-Sleep Scale (MOS-SS) (Double-Blind Phase)
Description: as for outcome 12
Time Frame: Week 19
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Pregabalin DB | Placebo
Number analyzed (Participants) | 147 | 147
participants | 67 | 60

14. Secondary Outcome: Weekly Mean Sleep Interference Score (Single-Blind Phase)
Description: Weekly mean sleep interference score was defined as the mean of the daily sleep interference diary ratings split into 7 day intervals. Participants rated how painful DPN has interfered with their sleep during the past 24 hours on an 11-point numeric rating scale ranging from 0 = does not interfere with sleep to 10 = completely interferes (unable to sleep due to pain). SB baseline refers to the last 7 pain diary entries up to and including Day 1.
Time Frame: SB Baseline, Week 1, 2, 3, 4, 5, 6
Population: SBAS included all participants who were enrolled into the single-blind treatment phase and received at least 1 dose of study treatment. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure and "n" signifies participants who were evaluable for specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin SB
Number analyzed (Participants) | 663
units on a scale
  SB Baseline (n= 663) | 5.9 (2.09)
  Week 1 (n= 657) | 5.1 (2.22)
  Week 2 (n= 636) | 4.5 (2.29)
  Week 3 (n= 614) | 4.1 (2.30)
  Week 4 (n= 589) | 3.8 (2.30)
  Week 5 (n= 566) | 3.7 (2.29)
  Week 6 (n= 548) | 3.6 (2.35)

15. Secondary Outcome: Weekly Mean Sleep Interference Score (Double-Blind Phase)
Description: Weekly mean sleep interference score was defined as the mean of the daily sleep interference diary ratings split into 7 day intervals. Participants rated how painful DPN has interfered with their sleep during the past 24 hours on an 11-point numeric rating scale ranging from 0 = does not interfere with sleep to 10 = completely interferes (unable to sleep due to pain).
Time Frame: DB Baseline, Week 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin DB | Placebo
Number analyzed (Participants) | 147 | 147
units on a scale
  DB Baseline (n= 147, 147) | 2.5 (1.79) | 2.3 (1.66)
  Week 7 (n= 144, 145) | 2.6 (1.92) | 2.7 (1.99)
  Week 8 (n= 143, 142) | 2.6 (1.98) | 3.0 (1.98)
  Week 9 (n= 140, 134) | 2.3 (1.88) | 2.7 (1.94)
  Week 10 (n= 138, 133) | 2.3 (1.90) | 2.7 (1.98)
  Week 11 (n= 138, 128) | 2.2 (1.81) | 2.5 (1.78)
  Week 12 (n= 136, 123) | 2.3 (1.90) | 2.4 (1.84)
  Week 13 (n= 134, 122) | 2.3 (1.87) | 2.3 (1.78)
  Week 14 (n= 133, 122) | 2.3 (1.93) | 2.3 (1.80)
  Week 15 (n= 132, 120) | 2.4 (1.93) | 2.3 (1.80)
  Week 16 (n= 132, 120) | 2.3 (1.90) | 2.3 (1.77)
  Week 17 (n= 129, 116) | 2.2 (1.88) | 2.2 (1.85)
  Week 18 (n= 128, 116) | 2.3 (1.92) | 2.3 (1.85)
  Week 19 (n= 121, 111) | 2.3 (2.05) | 2.2 (1.80)

16. Secondary Outcome: Endpoint Mean Sleep Interference Score (Single-Blind Phase)
Description: Endpoint mean sleep interference score was defined as the mean of the last 7 sleep interference diaries while receiving SB treatment. Participants rated how painful DPN has interfered with their sleep during the past 24 hours on an 11-point numeric rating scale ranging from 0 = does not interfere to 10 = completely interferes (unable to sleep due to pain).
Time Frame: Week 6
Population: SBAS included all participants who were enrolled into the single-blind treatment phase and received at least 1 dose of study treatment. Missing data were imputed using LOCF. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin SB
Number analyzed (Participants) | 658
units on a scale | 3.8 (2.42)

17. Secondary Outcome: Endpoint Mean Sleep Interference Score (Double-Blind Phase)
Description: Endpoint mean sleep interference score was defined as the mean of the last 7 sleep interference diaries while receiving DB treatment. Participants rated how painful DPN has interfered with their sleep during the past 24 hours on an 11-point numeric rating scale ranging from 0 = does not interfere to 10 = completely interferes (unable to sleep due to pain).
Time Frame: Week 19
Population: FAS included all participants randomized to double-blind treatment who received at least 1 dose of double-blind study treatment. Missing data were imputed using LOCF. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin DB | Placebo
Number analyzed (Participants) | 138 | 132
units on a scale | 2.4 (2.10) | 2.4 (2.05)

18. Secondary Outcome: Quality of Life Questionnaire- Diabetic Neuropathy (QOL-DN) (Single-Blind Phase)
Description: QOL-DN: 35-item participant-rated questionnaire used to assess impact of diabetic neuropathy on the quality of life of participants with diabetic neuropathy. Consists of 5 domains: Physical functioning(Ph Fn)/large fiber (sum of item 8, 11, 13-15, 24, 27-35; range -4 to 56); Activities of daily living (sum of item 12, 22, 23, 25, 26; range 0 to 20); Symptoms (sum of item 1-7, 9; range 0 to 32); Small fiber (sum of item 10, 16, 17, 18; range 0 to 16); Autonomic (sum of item 19, 20, 21; range 0 to 12) and total QOL score (sum of items 1-35) range: -4 to 136. Higher score implied worse QOL.
Time Frame: SB Baseline, Week 6
Population: SBAS included all participants who were enrolled into the single-blind treatment phase and received at least 1 dose of study treatment. Here "n" signifies participants who were evaluable for specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin SB
Number analyzed (Participants) | 665
units on a scale
  SB Baseline: Total QOL Scores (n= 665) | 42.6 (22.22)
  SB Baseline: Ph Fn/Large Fiber (n= 665) | 23.9 (13.07)
  SB Baseline: Activities of Daily Living (n= 665) | 3.2 (3.69)
  SB Baseline: Symptoms (n= 665) | 10.8 (5.55)
  SB Baseline: Small Fiber (n= 665) | 3.4 (3.40)
  SB Baseline: Autonomic (n= 665) | 1.3 (1.74)
  Week 6: Total QOL Scores (n= 618) | 29.3 (21.76)
  Week 6: Ph Fn/Large Fiber (n= 618) | 15.8 (12.62)
  Week 6: Activities of Daily Living (n= 618) | 2.2 (3.08)
  Week 6: Symptoms (n= 618) | 7.8 (5.72)
  Week 6: Small Fiber (n= 618) | 2.3 (2.99)
  Week 6: Autonomic (n= 618) | 1.1 (1.69)

19. Secondary Outcome: Quality of Life Questionnaire- Diabetic Neuropathy (QOL-DN) (Double-Blind Phase)
Description: as for outcome 18
Time Frame: Week 19
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin DB | Placebo
Number analyzed (Participants) | 138 | 134
units on a scale
  Total QOL Scores | 21.9 (20.02) | 24.1 (21.06)
  Ph Fn/Large Fiber | 11.4 (11.28) | 12.9 (12.72)
  Activities of Daily Living | 1.8 (2.85) | 1.8 (2.79)
  Symptoms | 6.1 (5.04) | 6.6 (5.29)
  Small Fiber | 1.8 (3.38) | 1.7 (2.50)
  Autonomic | 0.9 (1.55) | 1.1 (1.53)

20. Secondary Outcome: Pain Visual Analog Scale (VAS) (Single-Blind Phase)
Description: Participants rated their pain on a 100 millimeter (mm) Visual Analog Scale (VAS) ranging from 0 mm = no pain to 100 mm = worst possible pain.
Time Frame: SB Baseline, Week 6
Population: SBAS included all participants who were enrolled into the single-blind treatment phase and received at least 1 dose of study treatment. Here "n" signifies participants who were evaluable for specified time-point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Pregabalin SB
Number analyzed (Participants) | 665
mm
  SB Baseline (n= 665) | 68.1 (13.79)
  Week 6 (n= 621) | 39.8 (23.19)

21. Secondary Outcome: Pain Visual Analog Scale (VAS) (Double-Blind Phase)
Description: as for outcome 20
Time Frame: Week 19
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Pregabalin DB | Placebo
Number analyzed (Participants) | 138 | 134
mm | 25.3 (20.98) | 30.1 (23.44)

22. Secondary Outcome: Brief Pain Inventory-Short Form (BPI-sf) (Single-Blind Phase)
Description: BPI-sf: self-administered questionnaire developed to assess severity, impact of pain on daily functions, consisted of 5 questions. Questions 1-4 measured the severity of pain based on pain experienced over the past 24-hours on an 11-point scale ranged from 0 (no pain) to10 (worst possible pain). Question 5: 7 item subsets that measured level of interference of pain on daily functions on an 11-point scale ranged from 0 (does not interfere) to 10 (completely interferes).
Time Frame: SB Baseline, Week 6
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin SB
Number analyzed (Participants) | 665
units on a scale
  SB Baseline: Pain Severity (n= 665) | 6.1 (1.45)
  SB Baseline: Pain Interference (n= 665) | 5.2 (2.09)
  Week 6: Pain Severity (n= 637) | 3.9 (2.13)
  Week 6: Pain Interference (n= 637) | 3.1 (2.31)

23. Secondary Outcome: Brief Pain Inventory-Short Form (BPI-sf) (Double-Blind Phase)
Description: as for outcome 22
Time Frame: Week 19
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin DB | Placebo
Number analyzed (Participants) | 140 | 136
units on a scale
  Pain Severity | 2.6 (1.85) | 3.0 (2.03)
  Pain Interference | 2.0 (2.05) | 2.4 (2.10)

24. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) (Single-Blind Phase)
Description: HADS: self-administered questionnaire, consists of 2 sub-scales; measuring anxiety (HADS-A), and depression (HADS-D). Each sub-scale consists of 7 items on which participants responded as to how each item applies to them on a 4-point scale ranging from 0 (no anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score range for each sub-scale = 0 to 21, where higher score indicates more severe anxiety or depression.
Time Frame: SB Baseline, Week 6
Population: SBAS included all participants who were enrolled into the single-blind treatment phase and received at least 1 dose of study treatment. Here "N" (number of participants) signifies participants who were evaluable for this measure and "n" signifies participants who were evaluable for specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin SB
Number analyzed (Participants) | 663
units on a scale
  SB Baseline: HADS-A (n= 663) | 5.8 (3.95)
  SB Baseline: HADS-D (n= 663) | 5.3 (3.70)
  Week 6: HADS-A (n= 616) | 4.6 (3.54)
  Week 6: HADS-D (n= 616) | 4.0 (3.52)

25. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) (Double-Blind Phase)
Description: as for outcome 24
Time Frame: Week 19
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin DB | Placebo
Number analyzed (Participants) | 138 | 134
units on a scale
  HADS-A | 3.8 (2.94) | 4.3 (3.56)
  HADS-D | 3.3 (3.12) | 3.5 (3.28)

26. Secondary Outcome: Patient Global Evaluation of Study Medication (GESM) (Single-Blind Phase)
Description: GESM: single-item, self-administered treatment satisfaction questionnaire. Participants answered "how would you rate the study medication you received for pain?" on a 7-point scale ranging from 1 (very satisfied) to 7 (very dissatisfied). Number of participants in each category are reported.
Time Frame: Week 6
Population: SBAS included all participants who were enrolled into the single-blind treatment phase and received at least 1 dose of study treatment. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Pregabalin SB
Number analyzed (Participants) | 621
participants
  Very Satisfied | 241
  Somewhat Satisfied | 181
  Slightly Satisfied | 66
  Neither Satisfied Nor Dissatisfied | 71
  Slightly Dissatisfied | 22
  Somewhat Dissatisfied | 21
  Very Dissatisfied | 19

27. Secondary Outcome: Patient Global Evaluation of Study Medication (GESM) (Double-Blind Phase)
Description: as for outcome 26
Time Frame: Week 19
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Pregabalin DB | Placebo
Number analyzed (Participants) | 138 | 134
participants
  Very Satisfied | 80 | 64
  Somewhat Satisfied | 35 | 36
  Slightly Satisfied | 9 | 14
  Neither Satisfied Nor Dissatisfied | 6 | 10
  Slightly Dissatisfied | 5 | 2
  Somewhat Dissatisfied | 1 | 6
  Very Dissatisfied | 2 | 2

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin SB | Pregabalin DB | Placebo
Serious Adverse Events (participants affected / at risk) | 17/665 | 11/147 | 6/149
Other Adverse Events (participants affected / at risk) | 331/665 | 86/147 | 94/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin SB (N=665) | Pregabalin DB (N=147) | Placebo (N=149)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0
Generalised oedema (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Gangrene (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Tracheitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0
Burns first degree (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetic complication (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin SB (N=665) | Pregabalin DB (N=147) | Placebo (N=149)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Extrasystoles (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 2 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 3 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 5 | 0 | 2
Cataract (Eye disorders) | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 3 | 1 | 0
Cystoid macular oedema (Eye disorders) | 0 | 0 | 1
Diplopia (Eye disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 2 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 1 | 1 | 0
Retinal haemorrhage (Eye disorders) | 2 | 1 | 1
Retinal oedema (Eye disorders) | 0 | 0 | 1
Retinopathy hypertensive (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 12 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 1
Vitreous disorder (Eye disorders) | 1 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 15 | 2 | 3
Dental caries (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 15 | 5 | 6
Dry mouth (Gastrointestinal disorders) | 12 | 5 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 4 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 0
Lip disorder (Gastrointestinal disorders) | 1 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 22 | 4 | 5
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 2 | 4
Asthenia (General disorders) | 2 | 2 | 0
Breakthrough pain (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 4 | 1 | 0
Device breakage (General disorders) | 0 | 0 | 1
Face oedema (General disorders) | 1 | 1 | 0
Fatigue (General disorders) | 18 | 3 | 4
Feeling abnormal (General disorders) | 3 | 0 | 0
Feeling hot (General disorders) | 1 | 0 | 0
Feeling jittery (General disorders) | 1 | 0 | 0
Foaming at mouth (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 2 | 1 | 2
Generalised oedema (General disorders) | 2 | 1 | 1
Implant site pruritus (General disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 5 | 1 | 0
Irritability (General disorders) | 1 | 0 | 1
Local swelling (General disorders) | 1 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0
Oedema (General disorders) | 10 | 6 | 5
Oedema peripheral (General disorders) | 53 | 20 | 16
Pain (General disorders) | 1 | 2 | 1
Pyrexia (General disorders) | 1 | 0 | 0
Thirst (General disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0
Body tinea (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 3 | 3 | 0
Candidiasis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 5 | 4 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 2 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 3 | 1 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 1 | 0
Influenza (Infections and infestations) | 1 | 3 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 5 | 4 | 3
Oral herpes (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 1 | 0
Sinusitis (Infections and infestations) | 4 | 2 | 3
Skin candida (Infections and infestations) | 1 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 2
Tooth abscess (Infections and infestations) | 2 | 0 | 0
Tooth infection (Infections and infestations) | 3 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 11 | 7 | 7
Urinary tract infection (Infections and infestations) | 10 | 3 | 3
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 0
Ear canal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 2 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 3 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1 | 3
Limb injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 3 | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 2 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood amylase increased (Investigations) | 1 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 2
Blood glucose increased (Investigations) | 0 | 1 | 1
Blood pressure diastolic abnormal (Investigations) | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 2 | 0
Blood uric acid increased (Investigations) | 0 | 1 | 0
Body temperature increased (Investigations) | 1 | 0 | 0
Breath sounds abnormal (Investigations) | 1 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1
Haematocrit decreased (Investigations) | 1 | 0 | 0
Heart rate increased (Investigations) | 2 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1
Urinary casts (Investigations) | 0 | 0 | 1
Urine analysis abnormal (Investigations) | 1 | 0 | 1
Weight increased (Investigations) | 11 | 6 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 2
Fluid retention (Metabolism and nutrition disorders) | 2 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 5 | 0 | 2
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 3 | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 2 | 3
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Extremity contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 2 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 3 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 | 3 | 8
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Akathisia (Nervous system disorders) | 1 | 0 | 0
Allodynia (Nervous system disorders) | 3 | 2 | 2
Amnesia (Nervous system disorders) | 1 | 0 | 1
Areflexia (Nervous system disorders) | 2 | 0 | 1
Ataxia (Nervous system disorders) | 5 | 0 | 1
Balance disorder (Nervous system disorders) | 4 | 0 | 0
Burning sensation (Nervous system disorders) | 2 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular disorder (Nervous system disorders) | 1 | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 2 | 0 | 0
Coordination abnormal (Nervous system disorders) | 2 | 0 | 0
Decreased vibratory sense (Nervous system disorders) | 3 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 6 | 1 | 2
Disturbance in attention (Nervous system disorders) | 3 | 0 | 2
Dizziness (Nervous system disorders) | 45 | 4 | 2
Dizziness postural (Nervous system disorders) | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 29 | 4 | 4
Hyperaesthesia (Nervous system disorders) | 3 | 2 | 4
Hypersomnia (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 7 | 1 | 2
Lethargy (Nervous system disorders) | 2 | 1 | 1
Memory impairment (Nervous system disorders) | 3 | 0 | 0
Migraine (Nervous system disorders) | 2 | 0 | 1
Neuralgia (Nervous system disorders) | 2 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 3 | 1 | 1
Poor quality sleep (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Sedation (Nervous system disorders) | 5 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 2
Sinus headache (Nervous system disorders) | 1 | 1 | 0
Somnolence (Nervous system disorders) | 38 | 6 | 5
Tension headache (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 1
Agitation (Psychiatric disorders) | 2 | 0 | 0
Anorgasmia (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 0 | 0
Bradyphrenia (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 2 | 0 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 6 | 2 | 2
Depressive symptom (Psychiatric disorders) | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 2 | 0 | 0
Euphoric mood (Psychiatric disorders) | 1 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 11 | 0 | 2
Libido decreased (Psychiatric disorders) | 1 | 0 | 1
Mood swings (Psychiatric disorders) | 2 | 1 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 1
Nightmare (Psychiatric disorders) | 3 | 1 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 2 | 0 | 0
Thinking abnormal (Psychiatric disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1
Renal pain (Renal and urinary disorders) | 0 | 1 | 0
Urine odour abnormal (Renal and urinary disorders) | 1 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 3 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail hypertrophy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin tightness (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Hypertension (Vascular disorders) | 2 | 1 | 0
Hypotension (Vascular disorders) | 3 | 1 | 0
Intermittent claudication (Vascular disorders) | 0 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.